CLINICAL TRIAL: NCT03884270
Title: Self-Administered Hypnotherapy for Functional Dyspepsia
Brief Title: Functional Dyspepsia Hypnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Kinsinger (Other)
Responsible Party: Sponsor-Investigator, Sarah Kinsinger, Associate Professor of Medicine, Loyola University
Organization: Loyola University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 211673
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Results first posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-01

CONDITIONS: Functional Dyspepsia
Keywords: functional dyspepsia; hypnotherapy; functional gastrointestinal disorders
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: This is a non-randomized observational study designed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypnotherapy (Experimental): 7 sessions of on-line hypnotherapy treatment over the course of 12 weeks (1 new session every 2 weeks)
  Interventions: Behavioral: Hypnotherapy

INTERVENTIONS:
Behavioral: Hypnotherapy — 7 sessions of self-administered gut-directed hypnotherapy for functional dyspepsia

SUMMARY:
The purpose of this study is to evaluate the efficacy of a hypnotherapy treatment program for functional dyspepsia that can be self-administered using on-line audio recordings. This is a non-randomized study. All patients will receive 7 sessions of hypnotherapy treatment administered over a 12-week period.

The primary objective of the study is to determine the feasibility and acceptability of the self-administered hypnotherapy program. The secondary objective is to evaluate the effect of the treatment on participant reported symptom severity, quality of life, anxiety and depression.

DETAILED DESCRIPTION:
Functional dyspepsia (FD) is a very common health problem characterized by epigastric pain and/or postprandial fullness with no evidence of structural disease to explain the symptoms. There are few effective treatment options for FD, with medications having limited efficacy for the condition.

The goal of the current study is to test a 7-session hypnotherapy treatment specifically targeting symptoms of functional dyspepsia. The intervention will be provided via the Internet with pre-recorded audio files. In this trial, 23 adults diagnosed with functional dyspepsia in accordance with the Rome IV criteria will be included. Patients will meet with a licensed health psychologist for an initial study visit to determine their eligibility for hypnotherapy treatment. Following this screening visit, patients will receive an email with information for accessing the password-protected online platform where they will complete pre-treatment assessment forms and access treatment materials. Participants will complete baseline questionnaire data prior to beginning the hypnotherapy sessions and follow-up questionnaires at mid-treatment (6 weeks), post-treatment (12 weeks) and 3 months post-treatment. Participants will complete a new hypnotherapy session every 2 weeks over the course of 3 months and utilize a shorter, practice session 5 times per week.

The primary aim of the study is to assess feasibility and acceptability of the online treatment program by assessing the percentage of patients who log in to the web interface, utilize the materials sufficiently, complete the 12 week program, and report at least average satisfaction with the treatment. The secondary aim is to determine treatment effectiveness by measuring changes in pre- to post- treatment scores on a self-report functional dyspepsia symptom severity index (Patient Assessment of Upper Gastrointestinal Symptom Severity Index; PAGI-SYM). Additional endpoints include changes in pre- to post- treatment scores on a measure of disease-specific quality of life and psychological indices.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of functional dyspepsia by a gastroenterologist
2. Meeting ROME IV diagnostic criteria for functional dyspepsia
3. At least 18 yrs of age (no upper age limit)
4. Able to give informed consent
5. English speaking
6. Have daily personal access to the Internet via laptop or desktop computer, tablet or a smartphone.

Exclusion Criteria:

1. Concomitant organic gastrointestinal disease
2. Diagnosed or presenting with serious mental illness (e.g., eating disorder, schizophrenia, psychosis, obsessive-compulsive disorder, post-traumatic stress disorder, or a dissociative disorder)
3. Cognitive or language barriers that make completion of questionnaires difficult or limit understanding of a verbal intervention (hypnosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kinsinger, PhD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ford AC, Marwaha A, Sood R, Moayyedi P. Global prevalence of, and risk factors for, uninvestigated dyspepsia: a meta-analysis. Gut. 2015 Jul;64(7):1049-57. doi: 10.1136/gutjnl-2014-307843. Epub 2014 Aug 21. PMID 25147201
- [Background] Stanghellini V, Chan FK, Hasler WL, Malagelada JR, Suzuki H, Tack J, Talley NJ. Gastroduodenal Disorders. Gastroenterology. 2016 May;150(6):1380-92. doi: 10.1053/j.gastro.2016.02.011. PMID 27147122
- [Background] Ford AC, Forman D, Bailey AG, Axon AT, Moayyedi P. Initial poor quality of life and new onset of dyspepsia: results from a longitudinal 10-year follow-up study. Gut. 2007 Mar;56(3):321-7. doi: 10.1136/gut.2006.099846. Epub 2006 Aug 14. PMID 16908511
- [Background] Camilleri M, Stanghellini V. Current management strategies and emerging treatments for functional dyspepsia. Nat Rev Gastroenterol Hepatol. 2013 Mar;10(3):187-94. doi: 10.1038/nrgastro.2013.11. Epub 2013 Feb 5. PMID 23381190
- [Background] Palsson OS. Hypnosis Treatment of Gastrointestinal Disorders: A Comprehensive Review of the Empirical Evidence. Am J Clin Hypn. 2015 Oct;58(2):134-58. doi: 10.1080/00029157.2015.1039114. PMID 26264539
- [Background] Chiarioni G, Vantini I, De Iorio F, Benini L. Prokinetic effect of gut-oriented hypnosis on gastric emptying. Aliment Pharmacol Ther. 2006 Apr 15;23(8):1241-9. doi: 10.1111/j.1365-2036.2006.02881.x. PMID 16611286
- [Background] Calvert EL, Houghton LA, Cooper P, Morris J, Whorwell PJ. Long-term improvement in functional dyspepsia using hypnotherapy. Gastroenterology. 2002 Dec;123(6):1778-85. doi: 10.1053/gast.2002.37071. PMID 12454833
- [Background] Orive M, Barrio I, Orive VM, Matellanes B, Padierna JA, Cabriada J, Orive A, Escobar A, Quintana JM. A randomized controlled trial of a 10 week group psychotherapeutic treatment added to standard medical treatment in patients with functional dyspepsia. J Psychosom Res. 2015 Jun;78(6):563-8. doi: 10.1016/j.jpsychores.2015.03.003. Epub 2015 Mar 11. PMID 25791668
- [Background] Faramarzi M, Azadfallah P, Book HE, Rasolzadeh Tabatabai K, Taherim H, Kashifard M. The effect of psychotherapy in improving physical and psychiatric symptoms in patients with functional dyspepsia. Iran J Psychiatry. 2015;10(1):43-9. PMID 26005480
- [Background] Kawata H, Oka T. [The use of psychotropic drugs for functional gastrointestinal disorders: are they beneficial?]. Nihon Rinsho. 2012 Jan;70(1):84-8. Japanese. PMID 22413498
- [Background] Faramarzi M, Azadfallah P, Book HE, Tabatabaei KR, Taheri H, Shokri-shirvani J. A randomized controlled trial of brief psychoanalytic psychotherapy in patients with functional dyspepsia. Asian J Psychiatr. 2013 Jun;6(3):228-34. doi: 10.1016/j.ajp.2012.12.012. Epub 2013 Feb 15. PMID 23642981
- [Background] Jee SR, Jung HK, Min BH, Choi KD, Rhee PL, Kang YW, Lee SI; Korean Society of Neurogastroenterology and Motility. [Guidelines for the treatment of functional dyspepsia]. Korean J Gastroenterol. 2011 Feb;57(2):67-81. doi: 10.4166/kjg.2011.57.2.67. Korean. PMID 21350319
- [Background] Hjelland IE, Svebak S, Berstad A, Flatabo G, Hausken T. Breathing exercises with vagal biofeedback may benefit patients with functional dyspepsia. Scand J Gastroenterol. 2007 Sep;42(9):1054-62. doi: 10.1080/00365520701259208. PMID 17710670
- [Background] Haag S, Senf W, Tagay S, Langkafel M, Braun-Lang U, Pietsch A, Heuft G, Talley NJ, Holtmann G. Is there a benefit from intensified medical and psychological interventions in patients with functional dyspepsia not responding to conventional therapy? Aliment Pharmacol Ther. 2007 Apr 15;25(8):973-86. doi: 10.1111/j.1365-2036.2007.03277.x. PMID 17403002
- [Background] Hamilton J, Guthrie E, Creed F, Thompson D, Tomenson B, Bennett R, Moriarty K, Stephens W, Liston R. A randomized controlled trial of psychotherapy in patients with chronic functional dyspepsia. Gastroenterology. 2000 Sep;119(3):661-9. doi: 10.1053/gast.2000.16493. PMID 10982759
- [Background] Haug TT, Wilhelmsen I, Svebak S, Berstad A, Ursin H. Psychotherapy in functional dyspepsia. J Psychosom Res. 1994 Oct;38(7):735-44. doi: 10.1016/0022-3999(94)90026-4. PMID 7877128
- [Background] Arn I, Theorell T, Uvnas-Moberg K, Jonsson CO. Psychodrama group therapy for patients with functional gastrointestinal disorders--a controlled long-term follow-up study. Psychother Psychosom. 1989;51(3):113-9. doi: 10.1159/000288144. PMID 2636416
- [Background] Palsson OS, Turner MJ, Whitehead WE. Hypnosis home treatment for irritable bowel syndrome: a pilot study. Int J Clin Exp Hypn. 2006 Jan;54(1):85-99. doi: 10.1080/00207140500328666. PMID 16316885
- [Background] van Tilburg MA, Chitkara DK, Palsson OS, Turner M, Blois-Martin N, Ulshen M, Whitehead WE. Audio-recorded guided imagery treatment reduces functional abdominal pain in children: a pilot study. Pediatrics. 2009 Nov;124(5):e890-7. doi: 10.1542/peds.2009-0028. Epub 2009 Oct 12. PMID 19822590
- [Background] Stake-Nilsson K, Hultcrantz R, Unge P, Wengstrom Y. Complementary and alternative medicine used by persons with functional gastrointestinal disorders to alleviate symptom distress. J Clin Nurs. 2012 Mar;21(5-6):800-8. doi: 10.1111/j.1365-2702.2011.03985.x. Epub 2011 Dec 17. PMID 22175282
- [Background] Rutten JM, Vlieger AM, Frankenhuis C, George EK, Groeneweg M, Norbruis OF, Tjon a Ten W, Van Wering H, Dijkgraaf MG, Merkus MP, Benninga MA. Gut-directed hypnotherapy in children with irritable bowel syndrome or functional abdominal pain (syndrome): a randomized controlled trial on self exercises at home using CD versus individual therapy by qualified therapists. BMC Pediatr. 2014 Jun 4;14:140. doi: 10.1186/1471-2431-14-140. PMID 24894077
- [Background] Palsson OS. Standardized hypnosis treatment for irritable bowel syndrome: the North Carolina protocol. Int J Clin Exp Hypn. 2006 Jan;54(1):51-64. doi: 10.1080/00207140500322933. PMID 16316883
- [Background] Rentz AM, Kahrilas P, Stanghellini V, Tack J, Talley NJ, de la Loge C, Trudeau E, Dubois D, Revicki DA. Development and psychometric evaluation of the patient assessment of upper gastrointestinal symptom severity index (PAGI-SYM) in patients with upper gastrointestinal disorders. Qual Life Res. 2004 Dec;13(10):1737-49. doi: 10.1007/s11136-004-9567-x. PMID 15651544
- [Background] Talley NJ, Verlinden M, Jones M. Validity of a new quality of life scale for functional dyspepsia: a United States multicenter trial of the Nepean Dyspepsia Index. Am J Gastroenterol. 1999 Sep;94(9):2390-7. doi: 10.1111/j.1572-0241.1999.01363.x. PMID 10483997
- [Background] Talley NJ, Tack J, Ptak T, Gupta R, Giguere M. Itopride in functional dyspepsia: results of two phase III multicentre, randomised, double-blind, placebo-controlled trials. Gut. 2008 Jun;57(6):740-6. doi: 10.1136/gut.2007.132449. Epub 2007 Oct 26. PMID 17965059
- [Background] Talley NJ, Verlinden M, Jones M. Quality of life in functional dyspepsia: responsiveness of the Nepean Dyspepsia Index and development of a new 10-item short form. Aliment Pharmacol Ther. 2001 Feb;15(2):207-16. doi: 10.1046/j.1365-2036.2001.00900.x. PMID 11148439
- [Background] Labus JS, Mayer EA, Chang L, Bolus R, Naliboff BD. The central role of gastrointestinal-specific anxiety in irritable bowel syndrome: further validation of the visceral sensitivity index. Psychosom Med. 2007 Jan;69(1):89-98. doi: 10.1097/PSY.0b013e31802e2f24. PMID 17244851
- [Background] Derogatis LR, Melisaratos N. The Brief Symptom Inventory: an introductory report. Psychol Med. 1983 Aug;13(3):595-605. PMID 6622612

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypnotherapy
Started | 23
Completed | 22
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Participants enrolled in the study
Arm/Group | Hypnotherapy
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White/Caucasian | 17
  Non-Hispanic Black/African American | 3
  Hispanic (any race) | 2
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 23
Relationship status [Count of Participants; unit: Participants]
  Single | 7
  Committed relationship | 6
  Married | 10
Education [Count of Participants; unit: Participants]
  High school | 3
  Some college | 3
  Technical school or associates degree | 2
  Undergraduate degree | 8
  Some graduate school | 1
  Graduate degree | 6
Employment [Count of Participants; unit: Participants]
  Full-time | 15
  Part-time | 2
  Not working | 4
  Retired | 2
Prior mental health diagnosis [Count of Participants; unit: Participants] — Participants were asked to self report any current or past psychiatric diagnoses
  Participants
    Yes | 11
    No | 12
Functional dyspepsia Rome Criteria met [Count of Participants; unit: Participants] — The Rome IV Gastroduodenal disorders module was used to characterize participants as meeting postprandial distress syndrome and/or epigastric pain syndrome criteria
  Participants
    Postprandial distress syndrome only | 6
    Epigastric pain syndrome only | 2
    Postprandial distress syndrome and epigastric pain syndrome | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants That Complete the Hypnotherapy Program
Description: Feasibility will be calculated as the proportion of participants who complete the hypnotherapy treatment program in comparison to those who drop out before treatment is completed.
Time Frame: 12 weeks
Population: Participants enrolled in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Hypnotherapy
Number analyzed (Participants) | 23
Participants | 22

2. Primary Outcome: Treatment Satisfaction
Description: Treatment satisfaction will be assessed with a single item at the end of treatment asking how satisfied they were overall with their assigned treatment (on a 7-point scale from "Extremely dissatisfied" to "Extremely satisfied")
Time Frame: 12 weeks
Population: Participants enrolled in the study and completed 3-month follow-up surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Hypnotherapy
Number analyzed (Participants) | 22
Participants
  Extremely dissatisfied | 1
  Very dissatisfied | 0
  Somewhat dissatisfied | 0
  Neutral | 2
  Somewhat satisfied | 12
  Very satisfied | 4
  Extremely satisfied | 3

3. Primary Outcome: Satisfaction With Web Platform
Description: At the end of treatment, patients were asked an open-ended question to obtain feedback on their experience using the web-based platform for treatment. They were asked to rate their difficulty using the web platform on a 7-point scale from "Extremely difficult" to "Extremely easy".
Time Frame: 12 weeks
Population: Participants enrolled in the study and completed 3-month follow-up surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Hypnotherapy
Number analyzed (Participants) | 22
Participants
  Extremely easy | 17
  Moderately easy | 3
  Somewhat easy | 1
  Neutral | 1
  Somewhat difficult | 0
  Moderately difficult | 0
  Extremely difficult | 0

4. Secondary Outcome: The Patient Assessment of Upper Gastrointestinal Symptom Severity Index (PAGI-SYM) Will be Used to Assess Changes in Functional Dyspepsia Symptoms
Description: The PAGI-SYM is a 20-item self-report measure of functional dyspepsia symptom severity. The scale consists of 6 subscales (heartburn/regurgitation, nausea/vomiting, postprandial fullness/early satiety, bloating, upper abdominal pain, and lower abdominal pain). Each item is measured by a 6-point Likert scale ranging from 0 (no complaints) to 5 (severe complaints). Subscale scores are calculated by taking the mean of the items in each subscale. The total score is calculated by taking the mean of the subscale scores. Total scores range from 0 to 5, with higher scores indicating worse symptoms. The PAGI-SYM total score was regressed on the fixed effect of time period in a linear mixed effects regression model that included random intercepts to account for within-participant correlation. Least square mean differences were calculated as 3-month follow-up minus baseline.
Time Frame: Baseline, 3-months
Population: Participants enrolled in the study.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Hypnotherapy
Number analyzed (Participants) | 23
score on a scale | -0.82 (0.12)

5. Secondary Outcome: The Short Form Nepean Dyspepsia Index (NDI-SF) Will be Used to Assess Changes in Quality of Life Related to Functional Dyspepsia.
Description: The NDI-SF is a 10-item self-report disease specific quality of life questionnaire. The scale consists of 5 sub-scales (tension/anxiety, interference with daily activities, disruption to regular eating/drinking, knowledge towards/control over disease, interference with work/study). Each item is measured by a 5-point Likert scale ranging from 0 (not applicable) to 4 (extremely). Individual items are aggregated to obtain a total score ranging from 0 to 100 with higher scores indicating greater impairment in quality of life. The NDI-SF score was regressed on the fixed effect of time period in a linear mixed effects regression model that included random intercepts to account for within-participant correlation. Least square mean differences were calculated as 3-month follow-up minus baseline.
Time Frame: Baseline, 3 months
Population: Participants enrolled in the study.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Hypnotherapy
Number analyzed (Participants) | 23
score on a scale | -9.65 (1.75)

6. Secondary Outcome: The Visceral Anxiety Index (VSI) Will be Used to Assess Changes in Gastrointestinal Specific Anxiety.
Description: The VSI is a 15-item self-report questionnaire with responses ranging from 1 (strongly agree) to 6 (strongly disagree). The raw VSI score ranges from 0 (severe anxiety) to 75 (no anxiety). The VSI score was regressed on the fixed effect of time period in a linear mixed effects regression model that included random intercepts to account for within-participant correlation. Least square mean differences were calculated as 3-month follow-up minus baseline.
Time Frame: Baseline, 3 months
Population: Participants enrolled in the study.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Hypnotherapy
Number analyzed (Participants) | 23
score on a scale | 10.39 (2.73)

7. Secondary Outcome: The Brief Symptom Inventory (BSI) Will be Used to Assess Changes in Psychological Distress.
Description: The BSI is an 18-item self-report questionnaire with responses on a 5-point Likert scale, ranging from 0 (not bothered by a symptom at all) to 4 (extremely bothered). Three subscales are calculated (somatization, depression, and anxiety) and the subscales can be aggregated to calculate an overall global psychological distress score. The overall score and subscale scores are converted to T-scores (with a population mean of 50 and a standard deviation of 10). Higher T-scores indicate more psychological distress and T-scores ≥63 indicate clinically significant psychological distress. The BSI score was regressed on the fixed effect of time period in a linear mixed effects regression model that included random intercepts to account for within-participant correlation. Least square mean differences were calculated as 3-month follow-up minus baseline.
Time Frame: Baseline, 3 months
Population: Participants enrolled in the study
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Hypnotherapy
Number analyzed (Participants) | 23
score on a scale | -9.22 (1.34)

8. Secondary Outcome: Changes in Outpatient Physician Consultation Following Hypnotherapy Treatment.
Description: At both baseline and end of treatment, patients will be asked to report the number of outpatient visits and procedures they have had within the last 3 months related to their functional dyspepsia symptoms
Time Frame: Baseline, 12 weeks
Population: Participants enrolled in the study
Measure: Median (Inter-Quartile Range); unit: number of events
Arm/Group | Hypnotherapy
Number analyzed (Participants) | 23
number of events
  Number of outpatient visits at baseline | 2 [1 to 3]
  Number of outpatient visits at end of treatment | 1 [0 to 2]
  Number of procedures at baseline | 2 [1 to 2]
  Number of procedures at end of treatment | 1 [1 to 1]

9. Secondary Outcome: Number of Medications Used for Functional Dyspepsia
Description: At baseline and end of treatment, patients will be asked to report any medications they are taking related to their functional dyspepsia symptoms.
Time Frame: Baseline, 12 weeks
Population: Participants enrolled in the study
Measure: Median (Inter-Quartile Range); unit: number of medications
Arm/Group | Hypnotherapy
Number analyzed (Participants) | 23
number of medications
  Medications taking at baseline | 1 [1 to 2]
  Medications taking at end of treatment | 1 [1 to 2]

ADVERSE EVENTS:
Time Frame: 18 months
Description: We did not anticipate adverse events in this trial (there is no risk of serious adverse events, risk of all cause mortality, or other adverse events associated with GI hypnotherapy treatment); however, we did monitor for these while naturally tracking the patients for the study or through participant self-report.
Arm/Group | Hypnotherapy
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT03884270/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT03884270/ICF_001.pdf